CLINICAL TRIAL: NCT00527475
Title: Ranibizumab and Reduced Fluence Photodynamic Therapy for Choroidal Neovascularization in Age Related Macular Degeneration
Brief Title: Ranibizumab and Reduced Fluence PDT for AMD
Acronym: RAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Retina Associates (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAP AMD Trial
Record Dates: First submitted 2007-09-09; First posted 2007-09-11 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Macular Degeneration
Keywords: Anti-VEGF therapy; photodynamic therapy; neovascularization
MeSH Terms: conditions — Macular Degeneration; Neovascularization, Pathologic | interventions — Ranibizumab; Verteporfin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Active Comparator): Group I will receive 0.5 mg. ranibizumab intraocularly initially. This will be repeated monthly for 3 months total and then as needed over the period of one year.
  Interventions: Drug: ranibizumab
- Group II (Experimental): Group II will receive Reduced Fluence-PDT (25 Joules) followed by 0.5 mg. of ranibizumab intraocularly on the same day. The second group will receive the combination of ranibizumab and RF-PDT as needed over a period of one year.
  Interventions: Drug: ranibizumab; Drug: verteporfin

INTERVENTIONS:
Drug: ranibizumab — 0.5 mg. given as an intraocular injection
  Other Names: Lucentis
Drug: verteporfin — Standard dosage of 6 mgs. / meter2 of body surface area given intravenously.
  Other Names: Visudyne
  Arms: Group II

SUMMARY:
Single agent anti-VEGF therapies such as ranibizumab have shown great promise and have set the standard for visual outcomes in treating wet macular degeneration. However, they need to be administered frequently by intraocular injections with the attendant risk of endophthalmitis, lens damage, retinal detachment, and vitreous hemorrhage. The purpose of this trial is to see if using photodynamic therapy in combination with ranibizumab will decrease the number of treatments with ranibizumab.

DETAILED DESCRIPTION:
A randomized, prospective, multicenter trial will compare two groups of patients with subfoveal choroidal neovascularization secondary to AMD. One group will receive 0.5 mg. ranibizumab intraocularly initially. This will be repeated monthly for 3 months total and then as needed over the period of one year. The other group will receive Reduced Fluence-PDT (25 Joules) followed by 0.5 mg. of ranibizumab intraocularly on the same day. The second group will receive the combination of ranibizumab and RF-PDT as needed over a period of one year. Re-treatment will be determined by the individual investigator based on visual acuity, retinal thickness as measured by optical coherence tomography (OCT), and fluorescein angiography. Visual acuity and OCT measurements will be performed by masked examiners.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to sign informed consent.
2. Age greater than 50.
3. Evidence of macular degeneration in the form of drusen in either eye.
4. Visual acuity of 20/25 to 20/800.
5. Subfoveal choroidal neovascularization. Both occult and classic subtypes will be allowed. If lesion is purely occult there has to be one of the following:

   1. Recent loss of vision (5 letters on ETDRS or doubling of visual angle by snellen)
   2. Documented enlargement of lesion on FA
   3. Increase of 50 microns or more in the central subfield on OCT
   4. New blood
6. Total active lesion must be less than 12 disc areas in size. -

Exclusion Criteria:

1. Myopia, ocular histoplasmosis, or other retinal pathology that could affect vision
2. Previous treatment of the enrolled eye for CNV
3. Intraocular surgery within 6 weeks of enrollment
4. Geographic atrophy, subretinal fibrosis, or pigment epithelial tear involving the fovea of the eligible eye
5. Known hypersensitivity to verteporfin
6. Medical condition that would preclude regular follow-up for one year.
7. Previous vitrectomy
8. Media opacities limiting visual acuity, retinal examination, or retinal imaging.
9. A lesion where > 50% of the lesion is a pigment epithelial detachment. -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Callanan, MD, Study Chair — Texas Retina Associates
Locations (3):
- United States (3):
  - California Retina Consultants & Research Foundation, Santa Barbara, California
  - Associated Retinal Consultants, Ann Arbor, Michigan
  - Texas Retina Associates, Arlington, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab: Group I will receive 0.5 mg. ranibizumab intraocularly initially. This will be repeated monthly for 3 months total and then as needed over the period of one year.
- Reduced Fluence PDT & Ranibizumab: Group II will receive Reduced Fluence-PDT (25 Joules) followed by 0.5 mg. of ranibizumab intraocularly on the same day. The second group will receive the combination of ranibizumab and RF-PDT as needed over a period of one year.
Period: Overall Study
Arm/Group | Ranibizumab | Reduced Fluence PDT & Ranibizumab
Started | 30 | 30
Completed | 27 | 29
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Average age
  years | 79.1 (8.35) | 79.3 (7.23) | 79.2 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Less Than 15 Letters of ETDRS Visual Loss at 12 Months.
Time Frame: 1 year
Population: Fifty-six participants completed the full 12 month study. Four subjects did not return for the 12 month visit. No patients terminated the study due to adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Group I | Group II
Number analyzed (Participants) | 27 | 29
percentage of participants | 22 | 14

2. Secondary Outcome: Percentage of Participants With Retreatments Over One Year
Description: Number of days to retreatment outcome changed to frequency of retreatments at maintenance visits.
Time Frame: 1 year
Measure: Number; unit: % of subjects requiring additional injec
Arm/Group | Group I | Group II
Number analyzed (Participants) | 27 | 29
% of subjects requiring additional injec | 33 | 21

3. Secondary Outcome: Number of Injections Over 12 Months
Description: Additional number of ranibizumab injections given in each group over the 12 months
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Group I | Group II
Number analyzed (Participants) | 27 | 29
injections | 6.8 (2.49) | 3.0 (2.43)

4. Secondary Outcome: Percentage of Subjects Gaining More Than 15 ETDRS Letters of Acuity
Time Frame: 1 year
Measure: Number; unit: percentage
Arm/Group | Group I | Group II
Number analyzed (Participants) | 27 | 29
percentage | 33 | 31

5. Secondary Outcome: Improvement in OCT (Optical Coherent Tomography) Foveal Thickness at 12 Months
Description: Improvement in OCT (Optical coherent tomography) foveal thickness at 12 months/Number of microns in foveal thickness measurement
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Group I | Group II
Number analyzed (Participants) | 27 | 29
microns | 91.4 (12.8) | 104.1 (9.0)

ADVERSE EVENTS:
Arm/Group | Group I | Group II
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No